CLINICAL TRIAL: NCT01827293
Title: Promethazine vs. Lorazepam for Treatment of Vertigo in the Emergency Department: A Randomized Clinical Trial
Brief Title: Promethazine vs. Lorazepam for Treatment of Vertigo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shadi Asadollahi, Research Assistant, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB-067
Record Dates: First submitted 2013-04-02; First posted 2013-04-09 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Peripheral Vertigo.
MeSH Terms: conditions — Vertigo | interventions — Promethazine; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Promethazine (Active Comparator): IV promethazine (25 mg)
  Interventions: Drug: Promethazine; Drug: Lorazepam
- lorazepam (Active Comparator): IV lorazepam (2 mg)
  Interventions: Drug: Promethazine; Drug: Lorazepam

INTERVENTIONS:
Drug: Promethazine
Drug: Lorazepam

SUMMARY:
This study was a prospective, randomized, double-blind, parallel group clinical trial designed to compare the efficacy of intravenous (IV) promethazine and lorazepam for the treatment of peripheral vertigo in Emergency Department setting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Background history of positional vertigo

Exclusion Criteria:

* Unable to provide informed consent
* Pregnant or possibly pregnant
* Known allergy to study medications
* Use of antiemetic agents in the previous 24 hours
* Evidence of drug-induced vertigo or orthostatic hypotension
* Central pathologies/central origin for vertigo

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Mean change in vertigo intensity. | At 2 hours after intervention.
  The primary efficacy outcome was the mean change in the vertigo intensity score between pre- and post-intervention at 2 hours after administration of study medications.

SECONDARY OUTCOMES:
Efficacy and Safety outcome measures (nausea change-second dose-adverse events). | At 2-8 hours after intervention.
  Secondary outcomes included, mean change in nausea VAS score, need for second dose of study medications, and the rate of drug-related adverse events for the subjects in each study group after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Emam Hossein Hospital, Tehran, Nezam Abad, Iran